CLINICAL TRIAL: NCT01811940
Title: Multicenter Trial of Combined Pharmacotherapy to Treat Cocaine Dependence
Acronym: TACT2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6698; 1U01DA033310-01A1 (NIH)
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; adderall; topiramate
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adderall-ER and Topiramate (Experimental): Adderall-ER will be taken once per day in the morning or early afternoon since it may be activating. The dose is titrated to 60 mg per day or the maximum tolerated dose over two weeks and maintained for the duration of the study. Topiramate will be taken twice per day in the morning and the evening and titrated to 200mg/day or the maximum tolerated dose over the course of 6 weeks and maintained for the duration of the study.
  Interventions: Drug: Adderall-ER; Drug: Topiramate
- Placebo (Placebo Comparator): Placebo will be packaged in matching gelatin capsules similar to the pills in the active arm. Placebo will be taken as frequently and for the same duration as those taken in the active arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Adderall-ER — MAS-ER 60mg/day
  Other Names: Adderall extended release (MAS-ER)
  Arms: Adderall-ER and Topiramate
Drug: Topiramate — Topiramate 100 mg bid.
  Other Names: Topamax
  Arms: Adderall-ER and Topiramate
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The proposed protocol is a multi-site double-blind, placebo-controlled outpatient study of the safety and efficacy of Adderall-XR (MAS-ER) and topiramate in the treatment of cocaine dependence. 198 patients will be enrolled and 176 patients randomized in a 14-week trial. The proportion of participants achieving sustained cocaine abstinence for three consecutive weeks at the end of the study will be significantly greater for the combined pharmacotherapies group compared to the placebo group.

DETAILED DESCRIPTION:
The investigators hypothesize that the combination of an agent that increased baseline dopamine signaling (amphetamine) with one that reduced cocaine-induced dopamine release (topiramate) will improve dopamine regulation and be associated with improved cocaine use outcomes. 99 subjects at each of the two sites whom meet criteria for cocaine dependence, and all other study inclusion and exclusion criteria will be assigned to the 14-week double-blind, placebo-controlled treatment trial. Subjects will be randomized to receive either placebo or MAS-ER and topiramate. This proposal will test the hypothesis that MAS-ER and topiramate will promote cocaine abstinence. Participants who are randomized to the combination medication arm will have their dose titrated to 60 mg MAS-ER daily (over 2 weeks) and 200 mg topiramate a day (over 6 weeks) and maintained on this dose through week 13 of the trial. During week 14, participants will be tapered off both medications. All participants will receive a supportive behavioral treatment that emphasizes study procedure adherence. Starting in week one, all patients will receive incentives for compliance with study procedures on an escalating reinforcement schedule similar to that developed previously and not contingent on urine results. The purpose of the lead-out is to blind patients to the exact point of medication discontinuation and to provide naturalistic data on the effects of medication discontinuation. Moreover, a 3 month follow-up will be conducted to determine what happens to cocaine use after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-60 who meet DSM-IV criteria for cocaine dependence.
* Used cocaine at least 9 days in the past 28 days with at least weekly cocaine use.
* Able of giving informed consent and capable of complying with study procedures.

Exclusion Criteria:

* Meets DSM-IV-TR criteria for bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse.
* Individuals with any current Axis I psychiatric disorder as defined by DSM-IV-TR supported by the SCID-I/P that in the investigator's judgment are unstable, would be disrupted by study medication, or are likely to require pharmacotherapy or psychotherapy during the study period. Individuals who are currently stable on a psychotropic medication for at least 3 months may be included if in the investigator's opinion the psychotropic medication the patient is taking is compatible with the study medication (mixed amphetamine salts plus topiramate) and does not entail serious risk of adverse effects from the drug interactions. Individuals cannot be on any psychostimulants or other contraindicated medications.
* Individuals with a history of seizures or unexplained loss of consciousness
* History of allergic reaction to candidate medications (amphetamine or topiramate).
* Individuals with significant current suicidal risk.
* Women who are pregnant, nursing, or failure in sexually active female patients to use adequate contraceptive methods.
* Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (SBP > 140, DBP> 90,or HR > 100 when sitting quietly), acute hepatitis(patients with chronic mildly elevated transaminases < 3x upper limit of normal are acceptable), or uncontrolled diabetes.
* Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG, cardiac symptoms, fainting, open-heart surgery and/or arrhythmia, and family history of ventricular tachycardia/sudden death.
* Individuals with use of carbonic anhydrase inhibitors
* History of glaucoma
* History of kidney stones
* Use of drugs that may be additive to the bicarbonate lowering effects of topiramate
* Body Mass Index (BMI) < 18kg/m2
* History of failure to respond to a previous adequate trial of either of the candidate medications for cocaine dependence
* Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) which require medical intervention
* Individuals who are legally mandated (e.g., to avoid incarceration, monetary or other penalties,etc.) to participate in substance abuse treatment program
* Individuals with a current history (within the past 6 months) of amphetamine abuse or dependence including amphetamines such as methamphetamine and MDMA.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2013-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Levin, M.D., Principal Investigator — Columbia University; Kyle Kampman, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - STARS, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: stars website — http://stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 169 individuals enrolled in the trial and entered a 1 week placebo lead-in. 42 participants were not randomized due to several reasons including 16 being considered to be placebo-responders and 18 being lost to follow-up. 127 participants were then randomized.
Period: Overall Study
Arm/Group | Adderall-ER and Topiramate | Placebo
Started | 64 | 63
Completed | 42 | 37
Not Completed | 22 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adderall-ER and Topiramate | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (8.4) | 46.4 (8.4) | 46 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 47 | 49 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 52 | 52 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 42 | 81
  White | 11 | 10 | 21
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 6 | 6 | 12
education [Count of Participants; unit: Participants]
  High School or less | 38 | 41 | 79
  Some College | 14 | 13 | 27
  College or graduate school | 12 | 9 | 21
employment status [Count of Participants; unit: Participants]
  Full-time | 15 | 16 | 31
  Part-time | 7 | 6 | 13
  Unemployed/Other | 32 | 39 | 71
  not reported | 10 | 2 | 12
Currently married [Count of Participants; unit: Participants] | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Three Weeks of Cocaine Abstinence at End of Study
Description: The number of participants in each study arm achieving sustained cocaine abstinence for three consecutive weeks at the end of the study. This will be measured by self reported cocaine use on the daily Time line Follow Back (TLFB) and corroborated by the urine toxicology samples collected 3 times per week.
Time Frame: assessed during 14 weeks of trial, presented for last 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adderall-ER and Topiramate | Placebo
Number analyzed (Participants) | 64 | 63
Participants | 9 | 0

2. Secondary Outcome: Any Three Consecutive Weeks of Abstinence During Study
Description: The proportion of participants in each study arm achieving sustained cocaine abstinence for three consecutive weeks at any time during the 14 week trial. This will be measured by self reported cocaine use on the daily Time line Follow Back (TLFB)and corroborated by the urine toxicology samples collected 3 times per week.
Time Frame: 14 weeks of study or length of study participation
Measure: Count of Participants; unit: Participants
Arm/Group | Adderall-ER and Topiramate | Placebo
Number analyzed (Participants) | 64 | 63
Participants | 14 | 4

ADVERSE EVENTS:
Time Frame: collected during 14 weeks of trial or length of participation
Arm/Group | Adderall-ER and Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/64 | 2/63
Other Adverse Events (participants affected / at risk) | 52/64 | 44/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adderall-ER and Topiramate (N=64) | Placebo (N=63)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One patient was hospitalized for 48 hours due to an exacerbation of preexisting asthma. Upon receiving treatment, the symptoms subsided. Hospitalization was not considered related to study procedures.
inpatient rehabilitation (General disorders) | 1 (1) | 1 (1) — patient voluntarily entered an inpatient rehabilitation program.
leg swelling/pain (General disorders) | 0 (0) | 1 (1) — One participant presented to the ER with pain and swelling in both legs. He was admitted for 48 hours for observation in the hospital and treated with antibiotics.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adderall-ER and Topiramate (N=64) | Placebo (N=63)
headache (General disorders) | 9 (9) | 10 (10)
insomnia (General disorders) | 12 (12) | 6 (6)
URI (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9)
increased blood pressure (Cardiac disorders) | 10 (10) | 5 (5)
anorexia (Gastrointestinal disorders) | 9 (9) | 5 (5)
dry mouth (General disorders) | 10 (10) | 3 (3)
fatigue (General disorders) | 7 (7) | 6 (6)
GI upset (Gastrointestinal disorders) | 9 (9) | 3 (3)
muscle aches (General disorders) | 5 (5) | 7 (7)
paresthesia (General disorders) | 6 (6) | 5 (5)
anxiety (General disorders) | 6 (6) | 4 (4)
dizziness (General disorders) | 7 (7) | 3 (3)
drowsiness (General disorders) | 3 (3) | 7 (7)
diarrhea (Gastrointestinal disorders) | 5 (5) | 4 (4)
vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
increased heart rate (Cardiac disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT01811940/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT01811940/SAP_001.pdf